CLINICAL TRIAL: NCT04557254
Title: A Retrospective Single-center Comparative Analysis of Early and Long-term Results of Aortic Surgical Replacement Using Silver Acetate and Triclosan Impregnated Antimicrobial Grafts Versus Standard Dacron Vascular Grafts
Brief Title: Silver Acetate and Triclosan Antimicrobial Graft Evaluation for Surgical Repair of Aortic Disease
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Andrea Kahlberg, Principal Investigator, IRCCS San Raffaele
Other Study IDs: STAGER Study
Record Dates: First submitted 2020-09-08; First posted 2020-09-21 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Infective Graft Complications
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- silver-triclosan graft implantation (SynG group)
  Interventions: Device: graft
- standard Dacron graft implantation (DacrG group)
  Interventions: Device: graft

INTERVENTIONS:
Device: graft — evaluate the early and long-term clinical results, up to 5 years (through follow-up outpatient visits), of a silver and triclosan knitted collagen coated polyester vascular graft (InterGard Synergy), in patients submitted to aortic surgical repair, and compare them with concurrent results of standard Dacron grafts.

SUMMARY:
The number of surgical and endovascular aortic repairs is continuously increasing, and infective graft complications are observed more frequently. (1) Several etiopathogenetic factors may play a role in aortic prosthetic infections, including hematogenous seeding, local bacterial translocation, and iatrogenous contamination. Infectious graft complications represent a critical event requiring a multidisciplinary management. Knowledge on underlying microorganisms, antibiotic efficacy, risk factors, and prevention strategies has a key role in the management of this spectrum of infectious diseases involving the aorta.

the aim of the study is evaluate the early and long-term clinical results, up to 5 years (through follow-up outpatient visits), of a silver and triclosan knitted collagen coated polyester vascular graft (InterGard Synergy), in patients submitted to aortic surgical repair, and compare them with concurrent results of standard Dacron grafts. Results will be reported and analyzed according to the type of aortic disease requiring surgical repair.

ELIGIBILITY:
Inclusion Criteria:

• Patients submitted to aortic surgical repair (elective or emergent) with a silver and triclosan knitted collagen coated polyester vascular graft or standard Dacron grafts, for different aortic pathologies at the Division of Vascular Surgery, San Raffaele Scientific Institute, between 2012 and 2019

Exclusion Criteria:

• not present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have surgery aortic repair in which it was used a prosthesis containing antimicrobial agents or a standard vascular prosthesis (Dacron)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Number of patients without infectious complications | 30 days
  freedom from infectious complications (percentage)
Number of patients without infectious complications | 5 years
  freedom from infectious complications (percentage)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berard X, Stecken L, Pinaquy JB, Cazanave C, Puges M, Pereyre S, Bordenave L, M'Zali F. Comparison of the Antimicrobial Properties of Silver Impregnated Vascular Grafts with and without Triclosan. Eur J Vasc Endovasc Surg. 2016 Feb;51(2):285-92. doi: 10.1016/j.ejvs.2015.10.016. Epub 2015 Dec 9. PMID 26680451
- [Result] Kahlberg A, Melissano G, Tshomba Y, Leopardi M, Chiesa R. Strategies to treat thoracic aortitis and infected aortic grafts. J Cardiovasc Surg (Torino). 2015 Apr;56(2):269-80. Epub 2015 Jan 22. PMID 25608572
- [Derived] Kahlberg A, Bilman V, Bugna C, Rinaldi E, Mascia D, Loschi D, Chiesa R, Melissano G. Silver acetate and Triclosan Antimicrobial Graft Evaluation for surgical Repair of aortic disease (STAGER Study). Int Angiol. 2023 Oct;42(5):402-411. doi: 10.23736/S0392-9590.23.05101-5. Epub 2023 Nov 9. PMID 37943291